CLINICAL TRIAL: NCT05307445
Title: Treatment of Peri-Implant Mucositis With Standard of Care and Bioptron Hyperlight Therapy: A Parallel-Arm Clinical Trial
Brief Title: Treatment of Peri-Implant Mucositis With Standard of Care and Bioptron Hyperlight Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Gianna Maria Nardi, Clinical Professor, University of Roma La Sapienza
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 3464/23.12.2016
Record Dates: First submitted 2022-03-22; First posted 2022-04-01 (Actual); Last update posted 2022-04-01 (Actual); Status verified 2022-03

CONDITIONS: Mucositis Oral; Dental Implant Failed
Keywords: peri-implant mucositis; dental implants; Bioptron; photobiomodulation
MeSH Terms: conditions — Stomatitis | interventions — Low-Level Light Therapy

STUDY DESIGN:
Intervention Model Description: a randomised, double blind clinical trial
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- peri-implant mucositis treated with standard of care-professional mechanical debridement (Active Comparator): patients with peri-implant mucositis are treated with standard of care, i.e. professional mechanical debridement
  Interventions: Device: Photobiomodulation with Bioptron Hyperlight Therapy
- peri-implant mucositis treated with photobiomodulation in addition to standard treatment (Experimental): patients with peri-implant mucositis are treated with photobiomodulation in addition to standard treatment
  Interventions: Device: Photobiomodulation with Bioptron Hyperlight Therapy

INTERVENTIONS:
Device: Photobiomodulation with Bioptron Hyperlight Therapy — The Bioptron® Device provides polarized visible polychromatic noncoherent light with 90 W; light wavelength = 480-3400 nm; degree of polarization = 95%; specific power = 40 mW/cm2; energy density = 2.4 J/cm2. The duration of each treatment session was 10 min. Bioptron light was positioned 10 cm from the oral mucosa and a mouth opener was positioned for the entire duration of the session. Two weekly sessions during the first 4 weeks of treatment were applied.

SUMMARY:
Objectives:

The aim of this study was to evaluate in a cohort of patients with peri-implant mucositis: (a) the efficacy of professional mechanical debridement therapy assisted using Bioptron Hyperlight Therapy on the reduction of periodontal indexes (b) the reduction of total oxidative salivary stress.

Material and Methods Forty subjects with a diagnosis of peri-implant mucositis were enrolled in this study and randomly assigned to the study group (mechanical debridement therapy assisted using Bioptron Hyperlight Therapy) or control group (mechanical debridement therapy alone). The study duration was 6 months. Data on plaque index (PI), bleeding on probing (BoP), probing pocket depth (PPD) and pain relief on Visual Analogue Scale (VAS) were recorded at T0, T1 (14 days), T2 (1 month) and T3 (6 months). Group differences were assessed using Student's t-test and Pearson's Chi-squared test of homogeneity

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 30-60 years old.
* With diagnosis of peri-implant mucositis.
* Plaque index (PI) ≥ 40%.
* Al least one implant site with PPD≥4 mm, BOP+ and suppuration.
* No uncontrolled diabetes, cardiovascular diseases, bone metabolism disorders, no autoimmune diseases (lichen planus, pemphigoid, pemphigus and systemic lupus erythematosus).
* No pharmacological therapies, no chemo-radiotherapies.
* No smoking (>10 cigarettes/day), alcohol and/or drug consumption.
* No pregnancy or breastfeeding.
* No allergy.

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-01-07 (Actual); Primary Completion 2021-01-10 (Actual); Study Completion 2022-01-13 (Actual)

PRIMARY OUTCOMES:
Periodontal chart-Probing pocket depth (PPD) | Patients were assessed before study beginning (baseline)
  Probing pocket depth (PPD). PPD is a periodontal index. It is used to measure the depth of the tissue surrounding the dental implant; with notches measured in millimeters. The probe is placed in between the dental implant and gums and measures the depth of what is called the periodontal pocket- the space between the dental implant and the surrounding gums and bone.
Periodontal chart-Probing pocket depth (PPD) | Patients were assessed at 6 weeks (T1)
  Probing pocket depth (PPD). PPD is a periodontal index. It is used to measure the depth of the tissue surrounding the dental implant; with notches measured in millimeters. The probe is placed in between the dental implant and gums and measures the depth of what is called the periodontal pocket- the space between the dental implant and the surrounding gums and bone.
Periodontal chart-Probing pocket depth (PPD) | Patients were assessed at 12 weeks (T2)
  Probing pocket depth (PPD). PPD is a periodontal index. It is used to measure the depth of the tissue surrounding the dental implant; with notches measured in millimeters. The probe is placed in between the dental implant and gums and measures the depth of what is called the periodontal pocket- the space between the dental implant and the surrounding gums and bone.
Periodontal chart-Probing pocket depth (PPD) | Patients were assessed at 24 weeks (T3)
  Probing pocket depth (PPD). PPD is a periodontal index. It is used to measure the depth of the tissue surrounding the dental implant; with notches measured in millimeters. The probe is placed in between the dental implant and gums and measures the depth of what is called the periodontal pocket- the space between the dental implant and the surrounding gums and bone.
Periodontal chart-Bleeding on probing (BOP) | Patients were assessed before study beginning (baseline)
  Bleeding on probing (BOP). Bleeding on probing (BOP) is a parameter to measure soft tissue inflammation. It is measured with the use of a dental probe. The grading is :
  * 0: normal colour of gingiva, no inflammation, no bleeding;
  * 1: slight inflammation; no bleeding;
  * 2: moderate inflammation; presence of bleeding on probing;
  * 3: severe inflammation; tendency to spontaneus bleeding.
Periodontal chart-Bleeding on probing (BOP) | Patients were assessed at 6 weeks (T1)
  Bleeding on probing (BOP). Bleeding on probing (BOP) is a parameter to measure soft tissue inflammation. It is measured with the use of a dental probe. The grading is :
  * 0: normal colour of gingiva, no inflammation, no bleeding;
  * 1: slight inflammation; no bleeding;
  * 2: moderate inflammation; presence of bleeding on probing;
  * 3: severe inflammation; tendency to spontaneus bleeding.
Periodontal chart-Bleeding on probing (BOP) | Patients were assessed at 12 weeks (T2)
  Bleeding on probing (BOP). Bleeding on probing (BOP) is a parameter to measure soft tissue inflammation. It is measured with the use of a dental probe. The grading is :
  * 0: normal colour of gingiva, no inflammation, no bleeding;
  * 1: slight inflammation; no bleeding;
  * 2: moderate inflammation; presence of bleeding on probing;
  * 3: severe inflammation; tendency to spontaneus bleeding.
Periodontal chart-Bleeding on probing (BOP) | Patients were assessed at 24 weeks (T3)
  Bleeding on probing (BOP). Bleeding on probing (BOP) is a parameter to measure soft tissue inflammation. It is measured with the use of a dental probe. The grading is :
  * 0: normal colour of gingiva, no inflammation, no bleeding;
  * 1: slight inflammation; no bleeding;
  * 2: moderate inflammation; presence of bleeding on probing;
  * 3: severe inflammation; tendency to spontaneus bleeding.
Periodontal chart- Plaque index (PI) | Patients were assessed before study beginning (baseline)
  Plaque index (PI). Plaque index is used to evaluate the level and rate of plaque formation on dental implant surfaces. The grading is :
  * 0: no visible plaque;
  * 1: thin plaque layer detectable by scraping;
  * 2: moderate plaque layer; visible to the naked eye;
  * 3: abundant plaque layer.
Periodontal chart- Plaque index (PI) | Patients were assessed at 6 weeks (T1)
  Plaque index (PI). Plaque index is used to evaluate the level and rate of plaque formation on dental implant surfaces. The grading is :
  * 0: no visible plaque;
  * 1: thin plaque layer detectable by scraping;
  * 2: moderate plaque layer; visible to the naked eye;
  * 3: abundant plaque layer.
Periodontal chart- Plaque index (PI) | Patients were assessed at 12 weeks (T2)
  Plaque index (PI). Plaque index is used to evaluate the level and rate of plaque formation on dental implant surfaces. The grading is :
  * 0: no visible plaque;
  * 1: thin plaque layer detectable by scraping;
  * 2: moderate plaque layer; visible to the naked eye;
  * 3: abundant plaque layer.
Periodontal chart- Plaque index (PI) | Patients were assessed at 24 weeks (T3)
  Plaque index (PI). Plaque index is used to evaluate the level and rate of plaque formation on dental implant surfaces. The grading is :
  * 0: no visible plaque;
  * 1: thin plaque layer detectable by scraping;
  * 2: moderate plaque layer; visible to the naked eye;
  * 3: abundant plaque layer.

SECONDARY OUTCOMES:
Pain relief | Patients were assessed before study beginning (baseline)
  Pain relief assessed with the Numerical Rating Scale-11 (NRS-11)
Pain relief | Patients were assessed at 6 weeks (T1)
  Pain relief assessed with the Numerical Rating Scale-11 (NRS-11)
Pain relief | Patients were assessed at 12 weeks (T2)
  Pain relief assessed with the Numerical Rating Scale-11 (NRS-11)
Pain relief | Patients were assessed at 24 weeks (T3)
  Pain relief assessed with the Numerical Rating Scale-11 (NRS-11)

CONTACTS AND LOCATIONS:
Overall Officials: Roberto F Grassi, Prof, Study Director — University of Bari Aldo Moro
Locations (1):
- Roberto Felice Grassi, Bari, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nardi GM, Mazur M, Papa G, Petruzzi M, Grassi FR, Grassi R. Treatment of Peri-Implant Mucositis with Standard of Care and Bioptron Hyperlight Therapy: A Randomized Clinical Trial. Int J Environ Res Public Health. 2022 May 7;19(9):5682. doi: 10.3390/ijerph19095682. PMID 35565077